CLINICAL TRIAL: NCT05843253
Title: Phase 2 Study of Ribociclib-Containing Post-Radiotherapy Combinations in Pediatric and Young Adult Patients Newly Diagnosed With High-Grade Glioma, Including Diffuse Intrinsic Pontine Glioma: Ribociclib and Everolimus for HGG/DIPG Which Harbor Alterations of the Cell Cycle and/or PI3K/mTOR Pathways AND Ribociclib and Temozolomide for DHG, H3G34-mutant
Brief Title: Study of Ribociclib and Everolimus in HGG and DIPG or Ribociclib and Temozolomide in DHG, H3G34-mutant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT TarGeT-A; R01FD008167 (FDA)
Record Dates: First submitted 2023-04-20; First posted 2023-05-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-10

CONDITIONS: High Grade Glioma; Diffuse Intrinsic Pontine Glioma; Anaplastic Astrocytoma; Glioblastoma; Glioblastoma Multiforme; Diffuse Midline Glioma, H3 K27M-Mutant; Metastatic Brain Tumor; WHO Grade III Glioma; WHO Grade IV Glioma; Diffuse Hemispheric Glioma, H3 G34-Mutant
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma; Astrocytoma; Glioblastoma; Brain Neoplasms | interventions — ribociclib; Everolimus; Temozolomide

STUDY DESIGN:
Intervention Model Description: Ribociclib and Everolimus OR Ribociclib and Temozolomide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Stratum A (n=40) (Experimental): Patients with localized, intracranial, non-pontine, and non-thalamic HGG (who do not meet criteria for strata B, C, or D).
  Interventions: Drug: Ribociclib; Drug: Everolimus
- Stratum B (n=40) (Experimental): Patients with DIPG, defined as a tumor with pontine epicenter and diffuse involvement of at least 2/3 of the pons, with histopathology consistent with diffuse WHO grade 2-4 glioma (e.g., diffuse astrocytoma, anaplastic astrocytoma, glioblastoma, H3K27-altered diffuse midline glioma).
  Interventions: Drug: Ribociclib; Drug: Everolimus
- Stratum C (n=6-12) (Experimental): Patients with primary thalamic, spinal cord, and/or secondary (radiation-related) HGG.
  Interventions: Drug: Ribociclib; Drug: Everolimus
- Stratum D (n=6-12) (Experimental): Patients with metastatic/disseminated HGG, multifocal HGG, and/or gliomatosis cerebri who received craniospinal irradiation.
  Interventions: Drug: Ribociclib; Drug: Everolimus
- Stratum E (n=20) (Experimental): Patients with localized H3G34-mutant DHG
  Interventions: Drug: Ribociclib; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Ribociclib — Ribociclib PO qd on days 1-21
  Other Names: Kisqali
Drug: Everolimus — Everolimus PO qd on days 1-28
  Other Names: Afinitor
  Arms: Stratum A (n=40); Stratum B (n=40); Stratum C (n=6-12); Stratum D (n=6-12)
Drug: Temozolomide (TMZ) — Temozolomide PO qd on days 1-5 for the first 13 cycles
  Arms: Stratum E (n=20)

SUMMARY:
The goal of this study is to determine the efficacy of the 1) ribociclib and everolimus to treat pediatric and young adult patients newly diagnosed with a high-grade glioma (HGG), including DIPG, that have genetic changes in pathways (cell cycle, PI3K/mTOR) that these drugs target or 2) ribociclib and temozolomide to treat pediatric and young adult patients newly diagnosed with diffuse hemispheric glioma (DHG), H3G34-mutant.

The main question the study aims to answer is whether the combinations of ribociclib and everolimus or ribociclib and temozolomide can prolong the life of patients diagnosed with HGG/DIPG or DHG H3G34-mutant.

DETAILED DESCRIPTION:
This is a multicenter, international, phase 2 study of post-radiotherapy (RT) combination of ribociclib and everolimus to treat pediatric, adolescent, and young adult patients newly diagnosed with HGG and DIPG that harbor alterations of the cell cycle and/or PI3K/mTOR pathways to assess treatment efficacy (Stratum A-D Part 2). The study will include a feasibility cohort (Strata A-D, Part 1) to identify the dose of ribociclib PfOS (Powder for Oral Suspension) that is safe and tolerable in combination with everolimus. Efficacy for Strata A-D Part 2 study will be defined by progression-free survival (PFS; HGG [stratum A]) and Overall Survival (OS; DIPG [stratum B]), with key longitudinal biomarker correlatives. Outcomes among patients with primary thalamic, spinal cord, and/or secondary (radiation related) HGG (strata C) will be descriptively analyzed. Objective radiographic response rates and agent-specific toxicities will also be assessed, with a feasibility cohort to determine the recommended phase 2 dose (RP2D) of the combination of ribociclib and everolimus in patients with metastatic disease who received upfront craniospinal irradiation (stratum D).

The study was amended in October 2025 to also include an additional stratum, Stratum E, which will serve patients with localized DHG, H3G34-mutant with the combination of ribociclib and temozolomide. As most DHG, H3G34-mutant tumors are MGMT promoter methylated and receive temozolomide as part of standard of care, we are studying the adjuvant combination of ribociclib and temozolomide following upfront RT. Stratum E will open with a Phase 1 Run-In to determine the RP2D of ribociclib PfOS formulation in combination with temozolomide in patients newly-diagnosed with DHG, H3G34-mutant post-RT, with PK testing. Once the RP2D is determined, patients with localized DHG, H3G34-mutant will be enrolled on the Stratum E efficacy expansion cohort to descriptively assess survival outcomes, with similar longitudinal biomarker correlatives to the other strata.

Protocol therapy with the maintenance combination of either 1) ribociclib and everolimus or 2) ribociclib and temozolomide must begin no later than 35 calendar days post-completion of RT. The earliest patients can begin protocol treatment is 28 calendar days post-completion of RT. Each cycle will be 28 days in duration and treatment can continue up to a total of 26 cycles. For Strata A-D, Ribociclib will be given orally once daily for 3 weeks (days 1-21), with one week off. Everolimus will be given orally daily continuously (days 1-28). For Stratum E, Ribociclib will be given orally once daily for 3 weeks (days 1-21), and temozolomide will be given days 1-5 for the first 13 cycles (Year 1), and ribociclib alone will be given orally once daily for 3 weeks (days 1-21) for the subsequent 13 cycles (Year 2).

ELIGIBILITY:
TarGeT-A study strata definitions Part1: Initial Feasibility Study for the combination of ribociclib PfOS formulation with everolimus: Enrollment on this cohort will be limited to patients aged <21 years with primary intracranial localized HGG and DIPG

Part 2

* Stratum A: Patients with localized, intracranial, non-pontine, and non-thalamic HGG (who do not meet criteria for strata C-D)
* Stratum B: Patients with DIPG
* Stratum C: Patients with primary thalamic, spinal cord, and/or secondary/radiation-related HGG.
* Stratum D: Patients with metastatic/disseminated HGG, multifocal HGG, and/or gliomatosis cerebri who received CSI.

Stratum E

* Stratum E: Patients with localized DHG, H3G34-mutant.

Inclusion Criteria:

1. Inclusion criteria already met to enroll on TarGeT-SCR (central molecular and histopathologic screening) based on:

   1.1) Age: patients must be ≥12 months and ≤39 years of age at the time of enrollment on TarGeT-SCR. For the Part 1 Initial Feasibility Cohort (receiving ribociclib and everolimus) only: patients must be <21 years of age at the time of enrollment on this protocol.

   1.2) Diagnosis: patients with newly-diagnosed HGG, including DIPG are eligible. All patients must have histologic confirmation tumor tissue from diagnostic biopsy or resection, without exceptions. The diagnosis of HGG, including DIPG, must have been confirmed through TarGeT-SCR:
   * For the diagnosis of DIPG, patients must have a tumor with pontine epicenter and diffuse involvement of at least 2/3 of the pons, with histopathology, consistent with diffuse WHO grade 2-4 glioma
   * All other HGGs must be WHO grade 3 or 4.

   1.3) Disease status: There are no disease status requirements for enrollment
   * Patients without measurable disease are eligible.
   * Patients with metastatic or multifocal disease or gliomatosis cerebri who received upfront CSI are eligible
   * Patients with a primary spinal HGG are eligible
   * Patients with secondary, radiation-related HGG are eligible.
2. Inclusion criteria for assignment to TarGeT-A, for all strata:

2.1) Presence of at least one relevant actionable somatic alteration, detailed here:

* Pathogenic alterations presumed to cause activation of cell cycle:
* Amplification of CDK4 or CDK6
* Deletion of CDKN2A, CDKN2B, or CDKN2C
* Amplification of CCND1 or CCND2
* Pathogenic alterations presumed to cause activation of the PI3K/mTOR pathway:
* Deletion or mutation of PTEN
* Mutation or amplification of PIK3CA
* Mutation of PIK3R1
* Deletion or mutation of TSC1 or TSC2
* Patients with evidence of homozygous (biallelic) RB1 loss by sequencing are excluded from TarGeT-A
* Patients whose tumors harbor other alterations suspected to activate the cell cycle and/or PI3K/mTOR pathway could potentially also be eligible, but only following consensus recommendation by the international multidisciplinary molecular screening committee.
* For Stratum E: H3G34 (R/V) mutation

2.2) Performance Level: Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of ag. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

2.3) Prior Therapy for HGG:

* Surgery, RT, dexamethasone are permissible. Temozolomide administered concurrently with RT is permissible. Avastin/bevacizumab use is permitted given the last dose was administered > 21 days prior to enrollment. No other prior anticancer therapy for HGG will be allowed.
* Patients must have received photon or proton RT.
* Patients must have started RT < 42 calendar days from initial diagnosis defined as the date of diagnostic biopsy or resection. If a patient underwent 2 upfront surgeries (e.g., biopsy then resection or debulking), this is the date of the second surgery.
* RT delivered via photon or proton beam, must have been administered at a standard dose including (54 Gy in 30 fractions for DIPG, 54-59.4 Gy in 30-33 fractions), 45 Gy-54 Gy for primary spinal disease, and/or 36 Gy-39.6 Gy craniospinal for patients with spinal or leptomeningeal metastatic disease with supplemental boost to 45-54 Gy for metastasis within the thecal sac and 54 Gy-60 Gy for intracranial metastasis. Any variances in the radiotherapy dose within 10% of the standard doses outlined above will be discussed with the Sponsor-Investigator to confirm eligibility prior to study enrollment.
* Patients must enroll and start treatment No later than 35 calendar days post-completion of RT. The earliest patients can begin protocol treatment is 28 calendar days post-completion of RT.

2.4) Organ Function Requirements

2.4.1) Adequate Bone Marrow Function Defined as:

* Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3
* Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Hemoglobin >8 g/dL (may be transfused)

2.4.2) Adequate Renal Function Defined as:

* Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 OR
* Maximum serum creatinine based on (Schwartz et al. J. Peds, 106:522, 1985) age/gender as follows: 1 to < 2 years=0.6 mg/dL for males and females; 2 to < 6 years=0.8 mg/dL for males and females; 6 to < 10 years= 1.0 mg/dL for males and females; 10 to < 13 years=1.2 mg/dL for males and females. 13 to < 16 years=1.5 mg/dL for males and 1.4 mg/dL for females.

2.4.3) Adequate Liver Function Defined as:

* Total bilirubin must be ≤ 1.5 times institutional upper limit of normal for age
* AST(SGOT)/ALT(SGPT) ≤ 3 times institutional upper limit of normal
* Serum albumin ≥ 2g/dL

2.4.4) Adequate Cardiac Function Defined as:

* Ejection fraction of ≥ 50% by echocardiogram
* QTc ≤ 450 msec (by Bazett formula)

2.4.5) Adequate Neurologic Function Defined as: Patients with seizure disorder may be enrolled if well-controlled on anticonvulsants that are not strong inducers or inhibitors of CYP3A4/5.

2.4.6) Adequate Pulmonary Function Defined as: No evidence of dyspnea at rest, and a pulse oximetry >94% on room air if there is clinical indication for determination.

2.5) Ability to take medications by mouth: For ribociclib and everolimus strata, patients must be able to take study medications by mouth as administration via NG/NJ/G tube is not allowed.

2.6) Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines

2.7) Contraception: Male and female patients of childbearing potential must be willing to use a highly effective contraception method.

Exclusion Criteria

1. Pregnant or Breast-Feeding Pregnant or breast-feeding women will not be entered on this study due to known potential risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are post-menarchal. Patients of childbearing or child fathering potential must agree to use at least one highly effective method of contraception while being treated on this study and for 3 months after completing therapy. A woman is considered of childbearing potential if she is fertile, following menarche and until becoming post-menopausal unless permanently sterile. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient. A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy. Male participants should refrain from sperm donation throughout the duration of treatment and for 3 months after completion of therapy

   A highly effective contraception method is defined as one that results in a low failure rate (<1% per year) when used consistently and correctly. The following are considered highly effective contraception methods:
   * Combined estrogen and progesterone containing hormonal contraception associated with inhibition of ovulation.
   * Progesterone-only hormonal contraception associated with inhibition of ovulation.
   * Intra Uterine Device (IUD)
   * Intra Uterine hormone releasing system
   * Bilateral tubal occlusion
   * Vasectomized partner
   * Sexual abstinence (avoiding having heterosexual intercourse) The following contraceptive measures are NOT considered effective
   * Progesterone-only hormonal contraception (birth control pill) that that does NOT stop ovulation
   * Male or female condom with or without spermicide
   * Cap, diaphragm or sponge with spermicide
2. Concomitant Medications

   * Patients receiving corticosteroids are eligible. The use of corticosteroids must be reported.
   * Patients who are currently receiving another investigational drug are not eligible.
   * Patients who are currently receiving other anti-cancer agents are not eligible, with the exception of temozolomide given concurrently with RT only.
   * Patients who are receiving enzyme inducing anticonvulsants that are strong inducers or inhibitors of CYP3A4/5 are not eligible.
   * Patients who are receiving strong inducers or inhibitors of CYP3A4/5 are not eligible and should be avoided from 14 days prior to enrollment to the end of the study.
   * Patients who are receiving medications known to prolong QTc interval are not eligible.
   * Patients who are receiving therapeutic anticoagulation with warfarin or other coumadin-derived anticoagulants are not eligible. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed as long as the patient has adequate coagulation defined as aPTT < 1.5Xs ULN and INR < 1.5.
3. Patients who have an uncontrolled infection are not eligible.
4. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study are not eligible.
5. Patients with known clinically significant active malabsorption syndrome or other condition that could affect absorption are not eligible.
6. Patients with prior or ongoing clinically significant medical or psychiatric condition that, in the investigator's opinion, could affect the safety of the subject, or could impair the assessment of study results are not eligible.

Ages: 12 Months to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2034-08-28 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) in HGG (Part 2, Stratum A) | From date on treatment until date of Progressive Disease or death due to any cause or date of last follow-up, assessed up to 60 months
  To assess the efficacy of ribociclib and everolimus in pediatric and young adult patients newly diagnosed with HGG by estimating the distribution of PFS compared to molecularly-stratified and matched historical controls.
Overall Survival (OS) in DIPG (Part 2, Stratum B) | From date on treatment until date of death due to any cause or date of last follow-up, assessed up to 60 months
  To assess the efficacy of ribociclib and everolimus in pediatric and young adult patients newly diagnosed with DIPG by estimating the distribution of OS compared to molecularly-stratified and matched historical controls.
Establish MTD and RP2D of ribociclib and everolimus (Part 2, Stratum D) | Completion of Cycle 1 (28 days)
  To identify the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of the combination of ribociclib and everolimus given to patients with metastatic HGG who have received craniospinal irradiation CSI.
Number of participants with ribociclib and everolimus-related adverse events as assessed by CTCAE v5.0 (Part 1- initial feasibility study) | Completion of Cycle 1 (28 days)
  Identify the safe dose of ribociclib powder for oral solution (PfOS) formulation in combination with everolimus that is feasible in pediatric patients with newly-diagnosed HGG, including DIPG, with cell cycle and/or PI3K/mTOR pathway alterations. This will be achieved by calculating the number of participants with, as well as frequency and severity of, ribociclib and everolimus-related Adverse Events as assessed by CTCAE v5.0 in the first 6-12 patients enrolled
Establish RP2D of ribociclib and temozolomide (Phase 1 Run-In Stratum E) | Completion of Cycle 1 (28 days)
  Establish RP2D of ribociclib and temozolomide (Phase 1 Run-In Stratum E) Description: To identify the Recommended Phase 2 Dose (RP2D) of the combination of ribociclib and temozolomide given to patients with newly diagnosed localized DHG, H3G34-mutant who have received RT.

SECONDARY OUTCOMES:
Overall Survival in HGG | From date on treatment until date of death due to any cause or date of last follow-up, assessed up to 60 months
  Determine distribution of OS for pediatric and young adult patients newly-diagnosed with HGG which harbor cell cycle and/or PI3K/mTOR pathway alterations treated with post-RT ribociclib and everolimus.
Number of participants with ribociclib and everolimus-related adverse events as assessed by CTCAE v5.0 | From Day 1 of protocol treatment through 30 days following end of protocol treatment
  Assess and further characterize the safety and toxicity of post-RT combination of ribociclib and everolimus in pediatric and young adult patients newly diagnosed with HGG, including DIPG. This will be achieved by calculating the number of participants with, as well as frequency and severity of, ribociclib and everolimus-related Adverse Events as assessed by CTCAE v5.0.
Evaluate Health-Related Quality of Life Outcomes | At the end of every other Cycle (each cycle is 28 days)
  Evaluate health-related quality of life outcomes of pediatric and young adult patients newly-diagnosed with either 1) HGG, including DIPG, or 2) DHG, H3G34-mutant treated with combination of ribociclib and everolimus or ribociclib and temozolomide, by patient and/or parent reporting at key timepoints in therapy using the patient reported outcomes measurement information system (PROMIS) survey.
Overall Survival in DHG, H3G34-mutant | From date on treatment until date of death due to any cause or date of last follow-up, assessed up to 60 months
  Determine distribution of OS for pediatric and young adult patients newly-diagnosed with DHG, H3G34-mutant treated with post-RT ribociclib and temozolomide.
Number of participants with ribociclib and temozolomide-related adverse events as assessed by CTCAE v5.0 | From Day 1 of protocol treatment through 30 days following end of protocol treatment
  Assess and further characterize the safety and toxicity of post-RT combination of ribociclib and temozolomide in pediatric and young adult patients newly diagnosed with DHG, H3G34-mutant. This will be achieved by calculating the number of participants with, as well as frequency and severity of, ribociclib and temozolomide-related Adverse Events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Margot Lazow, MD, Study Chair — Nationwide Children's Hospital; Maryam Fouladi, MD, Principal Investigator — Nationwide Children's Hospital
Locations (21):
- United States (11):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Duke University Health System, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (2):
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Hopp Children's Cancer Center at NCT Heidelberg (KiTZ), Heidelberg, Baden-Wurttemberg, Germany
- Princess Máxima Center, Utrecht, Netherlands
- Starship Children's Hospital, Auckland, Grafton, New Zealand
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No